CLINICAL TRIAL: NCT04425135
Title: Phase II Single-arm Clinical Study of Camrelizumab Combined With Apatinib Mesylate and Standard Chemotherapy (Pemetrixed +Carboplatin) in Patients With Tyrosine Kinase Inhibitor Failure in ALK-positive Advanced NSCLC
Brief Title: Camrelizumab Combined With Apatinib Mesylate and Standard Chemotherapy (Pemetrixed + Carboplatin) in Patients With Tyrosine Kinase Inhibitor Failure in ALK-positive Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-ALKNSCLC-IIT-SHR1210-APA-C
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — camrelizumab; apatinib; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab +apatinib mesylate+Pemetrixed + Carboplatin (Experimental): Camrelizumab combined with apatinib mesylate,Pemetrixed and Carboplatin in the treatment（4-6 cycle）of effective (CR, PR, SD) patients continued to be treated with Camrelizumab combined with apadine mesylate until PD, toxicity intolerance, and other reasons that the researcher thinks need to stop the research treatment.
  Interventions: Drug: Camrelizumab; Drug: Apatinib; Drug: Pemetrixed; Drug: Carboplatin

INTERVENTIONS:
Drug: Camrelizumab — 200mg,D1,ivgtt, Q3w.
Drug: Apatinib — 250mg,Qd,Q3W.
Drug: Pemetrixed — 500 mg/m2,D1,ivgtt, Q3w.
Drug: Carboplatin — AUC=5~6,D1,ivgtt, Q3w.

SUMMARY:
This study is a phase II single-arm clinical study.The purpose of this study was to evaluate the efficacy and safety of carrelizumab combined with apatinib mesylate and standard chemotherapy (pemetrexed plus carboplatin) in patients with advanced non-squamous and non-small cell lung cancer who have failed tyrosine kinase inhibitor therapy and are ALK-positive.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 year，male or female；
* Subjects with histologically or cytologically confirmed advanced non-squamous non-small cell lung cancer, imaging stage IIIb~IV；
* ALK fusion gene is positive and meets the following conditions:

  1. First-line treatment failure after previous second-generation ALK-TKI (including but not limited to Aletinib, Ceritinib, Brigatinib, and x-396);
  2. Previous first-generation AlK-TKI (crizotinib) and second-generation ALK-TKI (including but not limited to Aletinib, Ceritinib, Brigatinib, and x-396) failed.
* Patients with at least one evaluable or measurable lesions as per RECIST version 1.1；
* Patients who have not previously received systematic chemotherapy for advanced lung cancer .Can also be enrolled if you have previously received Neoadjuvant or adjuvant therapy；
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1；
* Survival expectation ≥ 3 months;
* Women of childbearing age must have a serum pregnancy study within 2 weeks prior to the first dose and the results are negative. Female subjects of childbearing age and partners who are women of childbearing age must be contraceptive during the study period and within 180 days after the last administration of the study drug;
* The laboratory test value of the patient before medication should meet the following standards:

  1. Routine blood：WBC≥3.0 × 109/L；ANC≥1.5 × 109/L；PLT≥90 × 109/L；HGB≥9.0 g/dL；
  2. Liver function：TBIL≤1.5 × ULN，AST≤2.5 × ULN，ALT≤2.5 × ULN（Subjects with liver metastasis，AST≤5× ULN，ALT≤5 × ULN）；
  3. Renal function：Cr≤1.5 × ULN or CrCl ≥50 mL/min；
  4. Blood coagulation function：INR≤1.5，APTT≤1.5 ×ULN ；
* Subjects voluntarily joined the study, signed informed consent, good compliance, and followed up;

Exclusion Criteria:

* Tumor histology or cytology pathology confirmed that the components of small cell lung cancer or squamous cell carcinoma were more than 10%；
* Previously received any T cell costimulation or immunological checkpoint treatment, including but not limited to CTLA-4 inhibitors, PD-1 inhibitors, PD-L1/2 inhibitors or other T cell-targeting drugs；
* An active autoimmune disease requiring systemic treatment (such as the use of disease-alleviating drugs, corticosteroids or immunosuppressants) occurred within 2 years prior to the first administration.Alternative therapies (such as thyroxine, insulin or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic;
* Interstitial lung disease, drug-induced pneumonia, radiation pneumonitis requiring steroid therapy or active pneumonia with clinical symptoms or severe pulmonary dysfunction；
* Previous or current history of cancer other than NSCLC, except for non-melanoma skin cancer, in-situ cervical cancer or other cancers that have received curable treatment and have shown no signs of recurrence for at least 5 years；
* Has not fully recovered from toxicity and/or complications from any intervention prior to initiation of treatment (i.e., ≤ grade 1 or level required at baseline, excluding fatigue or hair loss);
* Have a tendency to hereditary bleeding or coagulopathy. Clinically significant bleeding symptoms or clear bleeding tendency within 3 months prior to enrollment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood++ and above；
* Patients with clear or suspected brain metastases. Patients with a history of brain metastases （must be completed and patients who are no longer in need of corticosteroid therapy） can be enrolled; for patients with asymptomatic, lesions ≤ 3 and single less than 10 mm, who is determined by the investigator whether or not to enroll ;
* There are clinical symptoms or diseases of the heart that are not well controlled, such as: (1) heart failure of NYHA class 2 or higher (2) unstable angina (3) myocardial infarction within 24 weeks (4) clinical need for treatment or Interventional supraventricular or ventricular arrhythmia；
* Uncontrolled hypertension after treatment (systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90mmHg), with a history of hypertensive crisis or hypertensive encephalopathy;Uncontrolled hyperglycemia after treatment (fasting glucose >8.9mmol/L);
* There is a clinically uncontrollable third interstitial fluid (such as pleural effusion/pericardial effusion, patients who do not need drainage or stop drainage for 3 days without significant increase in effusion can be enrolled)；
* Imaging (CT or MRI) shows that the tumor invades the large blood vessels or the investigator judges that the tumor is highly likely to invade the important blood vessels during the follow-up study and cause fatal bleeding.
* Have a history of immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency disease, or history of organ transplantation and bone marrow transplantation；
* Active hepatitis B (positive detection of hepatitis B virus surface antigen [HBsAg] in the screening period, and detection of HBV-DNA detection value higher than the upper limit of the normal value of the laboratory in the research center) or hepatitis C (in the screening period, hepatitis C virus surface antibody [ HCsAb] positive, HCV-RNA positive)；
* Subjects who have received or will receive live vaccine within 30 days of the first treatment；
* Subjects who simultaneously applied NMPA standard modern Traditional Chinese medicine preparation against lung cancer and immunomodulator;
* Allergic reactions to test drugs for this application；
* The investigator determined that the subject had other factors that might lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to approximately 1 year
  ORR, determined using RECIST v1.1, defined as best overall response (CR or PR) across all assessment time points during the period from enrolment to termination of trial treatment.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to approximately 1 year
  PFS, defined as the time from treatment to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | up to approximately 1 year
  Determined using RECIST v1.1 criteria
Overall Survival Rate at 1-year (OSR) | up to approximately 1 year

IPD SHARING:
Plan to Share IPD: Undecided